CLINICAL TRIAL: NCT04206176
Title: The Effects of loW Dose tIcagrelor on Platelet Function Testing in Patients With Stable Coronary arTery Disease: TWIST Trial
Brief Title: The Effects of loW Dose tIcagrelor on Platelet Function Testing in Patients With Stable Coronary arTery Disease
Acronym: TWIST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Naveen Seecheran, Principal Investigator, The University of The West Indies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CEC1152/06/19
Record Dates: First submitted 2019-11-28; First posted 2019-12-20 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Platelet Dysfunction Due to Drugs
Keywords: antiplatelet drugs; clopidogrel; ticagrelor; high on-treatment platelet reactivity; platelet function
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Intervention Model Description: Single, group crossover from clopidogrel to low dose ticagrelor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single group crossover (Experimental): The patients who are on a maintenance dose of clopidogrel 75mg once daily will be transitioned to ticagrelor 45mg twice daily after which they will be tested.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 45mg twice daily per oral administration
  Other Names: Low Dose Ticagrelor

SUMMARY:
This study aims to assess the effects of low dose ticagrelor on platelet function testing in patients with stable coronary artery disease.

DETAILED DESCRIPTION:
Dual antiplatelet therapy with aspirin and clopidogrel represents the standard of care for the prevention of recurrent ischemic events in patients undergoing percutaneous coronary intervention (PCI). For more than 20 years, dual antiplatelet therapy with aspirin and Clopidogrel has remained the cornerstone of treatment for patients with acute coronary syndrome (ACS). However, some patients have impaired clopidogrel response and thus persist with high on-treatment platelet reactivity (HPR) resulting in an increased risk of atherothrombotic events. The boxed warning added to the clopidogrel label underscoring the potential risk of adverse cardiovascular outcomes among patients with a "poor metabolizer" genotype and advocating the use of other antiplatelet medications or alternative dosing strategies for these patients has led to investigations of treatment options associated with more optimal platelet inhibition. These include switching to a novel generation P2Y12 inhibitor (e.g. prasugrel or ticagrelor).

Ticagrelor is an antagonist of the P2Y12 receptor. The drug was approved for use in the European Union by the European Medicines Agency on December 3, 2010. The drug was approved by the US Food and Drug Administration on July 20, 2011. The FDA indication for ticagrelor is a reduction of the rate of cardiovascular death, myocardial infarction (MI), and stroke in people with an acute coronary syndrome or history of myocardial infarction.

According to ESC 2017 guidelines, ticagrelor is the first-option treatment in patients with acute coronary syndrome with or without ST-segment elevation, irrespective of treatment strategy (invasive or non-invasive) - IB level of evidence. Furthermore, the 2017 ESC Focused Update on Duration of Dual Antiplatelet Therapy allows physicians to administer ticagrelor to patients with stable coronary artery disease undergoing percutaneous coronary intervention after taking thrombotic and hemorrhagic risk into consideration.

In healthy Chinese subjects, low-dose ticagrelor produced an antiplatelet efficacy similar to that of standard-dose ticagrelor, which was faster and more potent than the effect of clopidogrel. In the East Asian population, there is limited evidence available to date that compares low versus standard doses of ticagrelor to evaluate the clinical efficacy and safety. Larger and longer duration studies are warranted to more closely examine the appropriateness of lower doses of ticagrelor in this population.

The investigators postulate that inhibition of platelet aggregation in response to low dose Ticagrelor as opposed to the standard dose is non-inferior to that of Clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

1. between 18 and 74 years of age,
2. have stable coronary artery disease, already on DAPT with aspirin and clopidogrel for at least 6 months,
3. not on any physician-prescribed medications or complementary/alternative therapies,

Exclusion Criteria:

1. presence of active internal bleeding or history of bleeding diathesis or clinical findings associated with an increased risk of bleeding,
2. history of ischemic or hemorrhagic stroke, transient ischemic attack, intracranial neoplasm, arteriovenous malformation, or aneurysm,
3. history of clinical and/or hemodynamic instability,
4. within 1 month of placement of a bare-metal stent,
5. within 30 days of coronary artery bypass graft surgery or PCI without a stent placed,
6. planned coronary revascularization,
7. treatment with fibrin-specific fibrinolytic therapy <24 h or non-fibrin-specific fibrinolytic therapy <48 h,
8. use of an oral anticoagulation agent or international normalized ratio >1.5,
9. body weight <60 kg,
10. age >75 years,
11. hemoglobin <10 g/dL,
12. platelet count <100×106/μL,
13. creatinine >2 mg/dL,
14. hepatic enzymes >2.5 times the upper limit of normal,
15. pregnancy and/or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical effectiveness and safety of low ticagrelor as compared to standard dose clopidogrel based on platelet reaction units (PRU). | 2 weeks
  Platelet Reaction Units of low dose ticagrelor vs. standard dose clopidogrel

CONTACTS AND LOCATIONS:
Locations (1):
- The University of the West Indies, Saint Augustine, North, Trinidad and Tobago

REFERENCES:
- [Derived] Seecheran N, Boodhai B, Maharaj A, Ramdeen A, Debideen N, Ochalal V, Singh R, Seecheran R, Seecheran V, Persad S, Abdullah H, Peram L, Motilal S, Tello-Montoliu A, Schneider D. The Effect of Low-Dose Ticagrelor on Platelet Function Profiles in Patients With Stable Coronary Artery Disease in Trinidad: The TWIST Pilot Study. Cardiol Ther. 2020 Dec;9(2):493-503. doi: 10.1007/s40119-020-00195-2. Epub 2020 Aug 6. PMID 32766961